CLINICAL TRIAL: NCT06899360
Title: Evaluation of Clinical Progression, Prognostic Factors, and Quality of Life in Patients with Age-related Macular Degeneration (VERA-nAMD).
Brief Title: Evaluation of Clinical Progression, Prognostic Factors, and Quality of Life in Patients with Age-related Macular Degeneration.
Acronym: VERA-AMD
Status: Recruiting | Type: Observational
Sponsor: University of Udine (Other)
Responsible Party: Principal Investigator, Daniele Veritti, Prof., University of Udine
Other Study IDs: OCU_DMED_2025_1
Record Dates: First submitted 2025-03-12; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Age-Related Macular Degeneration
Keywords: age-related macular degeneration; artificial intelligence; anti-VEGF
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational cohort of patients with age-related macular degeneration: Observational cohort of patients with age-related macular degeneration eventually receiving anti-VEGF agents as per clinical practice.

SUMMARY:
The VERA-AMD study is a prospective, observational study designed to evaluate clinical progression, prognostic factors, and quality of life in patients with age-related macular degeneration (AMD). The study aims to analyze real-world clinical data to identify key predictors of disease progression and functional outcomes, with the goal of optimizing AMD management. The study involves 200 patients aged ≥50 with a confirmed diagnosis of AMD, monitored through routine clinical practice. Primary outcomes include progression rates to advanced AMD and changes in visual acuity, while secondary outcomes focus on retinal morphology and quality of life. Anti-VEGF therapy and AI-based fluid analysis will be integrated to explore their impact on disease progression and patient outcomes.

DETAILED DESCRIPTION:
The VERA-AMD study is a prospective, non-interventional, observational study investigating the clinical course, prognostic factors, and quality of life in patients with age-related macular degeneration (AMD). AMD is a leading cause of vision loss among the elderly, manifesting as either neovascular ("wet") AMD (nAMD) or geographic atrophy ("dry") AMD (GA-AMD). Despite advances in treatment, there is considerable variability in disease progression and response to therapy. This study aims to fill this gap by analyzing real-world data to identify predictors of disease progression and functional outcomes, ultimately improving clinical management strategies.

Study Objectives

The study's main objectives are to:

Assess the clinical progression of AMD in routine clinical practice. Identify prognostic factors associated with favorable or unfavorable disease outcomes.

Evaluate the impact of AMD on patient quality of life using validated questionnaires.

Methodology

Design: Prospective, non-profit, observational study. Population: 200 patients aged ≥50 years with confirmed AMD in at least one eye. Inclusion Criteria: Confirmed diagnosis of AMD, scheduled follow-up according to clinical practice.

Exclusion Criteria: Significant ocular or systemic diseases affecting visual outcomes.

Outcomes

Primary Outcome: Progression rate to advanced AMD, expressed as cases per 100 patient-years.

Secondary Outcomes: Changes in visual acuity, retinal morphology assessed by optical coherence tomography (OCT), and patient-reported quality of life.

Anti-VEGF Therapy and AI-Based Fluid Analysis

A significant part of the study focuses on the role of anti-VEGF treatment in controlling disease progression, especially in nAMD. Anti-VEGF agents such as aflibercept and ranibizumab are standard treatments for neovascular AMD, aiming to reduce fluid accumulation and neovascularization. The study will explore the relationship between treatment regimens (fixed vs. as-needed dosing) and clinical outcomes, including visual acuity and anatomical changes.

Artificial intelligence (AI)-based analysis of retinal fluid dynamics will be employed using OCT imaging data. Machine learning algorithms will be applied to identify patterns in fluid accumulation and disease progression, improving early detection and personalized treatment approaches.

Data Collection and Statistical Analysis

Data will be collected through regular clinical visits, OCT imaging, and visual acuity testing. Statistical analysis will include repeated measures models to evaluate disease progression and predictors of clinical outcomes. Sample size calculations anticipate a 5.2% annual progression rate in early/intermediate AMD and a 19.7% rate in advanced AMD, with an 80% statistical power at a 0.05 significance level.

Timeline

Interim analysis after 12 months (50 patients with follow-up). Primary analysis after 12 months (all patients). Follow-up analysis at 36 months. Consent and Ethics

Informed consent will be obtained from all participants. Data will be anonymized and handled according to ethical guidelines and institutional review board (IRB) protocols.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 50 years.
* confirmed diagnosis of AMD in at least one eye.
* follow-up scheduled according to standard clinical practice.

Exclusion Criteria:

* presence of other significant ocular conditions that could affect visual acuity.
* systemic conditions that make the patient unsuitable for long-term follow-up.

Ages: 50 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by age-related macular degeneration
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Best-corrected visual acuity (BCVA) | through study completion, 36 months
  visual acuity measured as ETDRS letters

SECONDARY OUTCOMES:
Self-reported vision-targeted quality of life | through study completion, 36 months
  Self-reported vision-targeted quality of life will be measured using National Eye Institute Visual Functioning Questionnaire 25 (VFQ-25). [Score 0-100, higher scores mean a better outcome]
Fluid volume (nL) in the retinal compartments | through study completion, 36 months
  Artificial intelligence based fluid analysis. Measurement of fluid volume (nL) in the intraretinal, subretinal and sub retinal pigment epithelium compartments
central retinal thickness | through study completion, 36 months
  central retinal thickness

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Veritti, Principal Investigator — Department of Ophthalmology, University of Udine
Locations (1):
- Department of Ophthalmology, Udine, UD, Italy

IPD SHARING:
Plan to Share IPD: Undecided